CLINICAL TRIAL: NCT00422448
Title: BRAF and Nevi.Nevi Are Common Benign Pigmented Tumors of the Skin. Mutations in So-called BRAF and NRAS Genes Genes Appear to be Initiating Events Responsible for the Formation of Nevi.
Brief Title: Study to Test Genetic Alterations Among Different Dermoscopic Types of Melanocytic Nevi.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Department of Dermatology, Medical University of Graz Austria, Iris Zalaudek
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: V9-B05 (FWF)
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Results first posted 2011-01-14 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2010-12

CONDITIONS: Nevi
Keywords: Dermoscopy; Histopathology; Genetics; Nevi; Nevogenesis
MeSH Terms: conditions — Nevus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nevi from participants (Experimental): Benign nevi dermoscopically sub-classified into 4 dermoscopic types (i.e., with globular, reticular, mixed pattern with globules in the center and mixed pattern with globules at the periphery) were excised from healthy volunteers for further genetical analysis
  Interventions: Genetic: To test the frequency of BRAF and NRAS mutations among nevi

INTERVENTIONS:
Genetic: To test the frequency of BRAF and NRAS mutations among nevi — Benign nevi excised for the study purpose where genetically analyzed for the presence/absence of BRAF and NRAS mutations
  Other Names: NM_004333; Homo sapiens v-raf murine sarcoma viral oncogene homolog B1

SUMMARY:
This project is a multicenter study in which we will investigate a dual concept of nevogenesis. Study location is the Department of Dermatology at the Medical University of Graz in collaboration with centers in Austria (Vienna), Italy (Naples, Benevento, Modena), Spain (Barcelona) and the United States (New York).

The hypothesis is that small congenital melanocytic nevi (CMN), "early" acquired melanocytic nevi in childhood (AMN) and dermal nevi, all dermatoscopically characterized by globular pattern, belong to the same spectrum of genetically determined melanocytic proliferations that develop due to endogenous pathways, in contrast to "true" acquired melanocytic nevi, dermatoscopically showing reticular pattern, that develop due to exogeneous factors such as UV-exposure.

DETAILED DESCRIPTION:
The investigations to this study will verify whether small CMN, "early" AMN and dermal nevi, characterized by globular pattern differ in their genetic alterations compared to reticular typed nevi. It will be expected that globular typed nevi and eventually dermal nevi lack B-RAF mutations whereas reticular nevi show alterations in the B-RAF gene. Study location: Graz

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 9 to 80 years showing one or more dermoscopically benign nevi with either uniform globular-cobblestone pattern or reticular pattern or a combination of both types

Exclusion Criteria:

* Children under the age of 9 years
* Pregnant woman
* Patients with atypical nevi (i.e., melanoma cannot be clinically ruled out)
* Patients with immunosuppression
* Patients with sun exposure 4 weeks before enrollment

Ages: 9 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-09; Primary Completion 2009-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Zalaudek, MD, Study Chair — Department of Dermatology, Medical University of Graz
Locations (1):
- Department of Dermatology, Medical University of Graz, Graz, Austria

REFERENCES:
- [Background] Zalaudek I, Grinschgl S, Argenziano G, Marghoob AA, Blum A, Richtig E, Wolf IH, Fink-Puches R, Kerl H, Soyer HP, Hofmann-Wellenhof R. Age-related prevalence of dermoscopy patterns in acquired melanocytic naevi. Br J Dermatol. 2006 Feb;154(2):299-304. doi: 10.1111/j.1365-2133.2005.06973.x. PMID 16433800
- [Background] Zalaudek I, Hofmann-Wellenhof R, Soyer HP, Ferrara G, Argenziano G. Naevogenesis: new thoughts based on dermoscopy. Br J Dermatol. 2006 Apr;154(4):793-4. doi: 10.1111/j.1365-2133.2006.07152.x. No abstract available. PMID 16536840
- [Derived] Pellacani G, Scope A, Ferrari B, Pupelli G, Bassoli S, Longo C, Cesinaro AM, Argenziano G, Hofmann-Wellenhof R, Malvehy J, Marghoob AA, Puig S, Seidenari S, Soyer HP, Zalaudek I. New insights into nevogenesis: in vivo characterization and follow-up of melanocytic nevi by reflectance confocal microscopy. J Am Acad Dermatol. 2009 Dec;61(6):1001-13. doi: 10.1016/j.jaad.2009.04.018. Epub 2009 Oct 14. PMID 19833408
- See also: Webpage of the sponsoring organization — http://www.fwf.ac.at/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pigmented lesion clinic from October 2006 to March 2009
Pre-assignment Details: Insufficient prospective accrual of patients during the 1st year of enrollment lead to additional retrospective inclusion of a dataset of 21 paraffin-embedded tissue specimens from excised nevi .
Groups:
- Nevi: with or without BRAF and NRAS
Period: Overall Study
Arm/Group | Nevi
Started | 43 (22 prospectively enrolled during study period and 21 retrospectively enrolled)
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nevi
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.3 (9.413)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 20
Region of Enrollment [Number; unit: participants]
  Austria | 22
  Italy | 21

OUTCOME MEASURES:

1. Primary Outcome: Frequency of BRAF Mutations Among Nevi
Description: All nevi were analyzed for BRAF mutations using the (less sensitive) Sanger method. A random subset of nevi was also analyzed using the (more sensitive) Ultradeep pyro-sequencing method (UDPS). The frequency is reported here as the number of BRAF mutations found by each method.
Time Frame: up to 30 months
Population: All nevi were analyzed for BRAF mutations using the (less sensitive) Sanger method. A random subset of nevi was also analyzed using the (more sensitive) Ultradeep pyro-sequencing method (UDPS). The frequency is reported here as the number of BRAF mutations found by each method.
Measure: Number; unit: BRAF mutations
Units Other Than Participants: nevi
Arm/Group | Nevi
Number analyzed (Participants) | 43
Number analyzed (nevi) | 45
BRAF mutations
  Sanger method (n=45) | 6
  UDPS (n=24) | 19

2. Secondary Outcome: Frequency of NRAS Mutations Among Nevi
Description: All nevi were analyzed for NRAS mutations using the (less sensitive) Sanger method. The (more sensitive) Ultradeep pyro-sequencing method (UDPS) is not applicable for this mutation. The frequency is reported here as the number of NRAS mutations from the analyzed nevi.
Time Frame: 30 months
Population: All nevi were analyzed for NRAS mutations using the (less sensitive) Sanger method. The (more sensitive) Ultradeep pyro-sequencing method (UDPS) is not applicable for this mutation. The frequency is reported here as the number of NRAS mutations from the analyzed nevi.
Measure: Number; unit: NRAS mutations
Units Other Than Participants: number of nevi
Arm/Group | Nevi
Number analyzed (Participants) | 43
Number analyzed (number of nevi) | 45
NRAS mutations | 0

ADVERSE EVENTS:
Time Frame: were not collected or assessed
Description: postoperative complications were not collected or assessed
Arm/Group | Nevi
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
During first year of enrollment too few patients agreed to participate. Therefore a sample of 21 nevi were additionally retrospectively included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No